CLINICAL TRIAL: NCT03449238
Title: Pembrolizumab And Stereotactic Radiosurgery (Srs) Of Selected Brain Metastases In Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1710018694
Record Dates: First submitted 2018-02-14; First posted 2018-02-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients with metastatic breast cancer with at least 2 brain metastases, eligible to receive SRS. Patients will complete radiation therapy within 1 week and Pembrolizumab may be continued every 3 weeks until evidence of brain progression or serious adverse toxicity. Patients will be followed until death.
  Pembrolizumab infusion will be given on Day 4 (+/-1) after SRS treatment at the standard dose of 200mg IV over 30 minutes and repeated every 3 weeks until disease progression or unacceptable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and SRS (Other): Pembrolizumab infusion will be given on Day 4 (+/-1) after SRS treatment at the standard dose of 200mg IV over 30 minutes and repeated every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab infusion will be given on Day 4 (+/-1) after SRS treatment at the standard dose of 200mg IV over 30 minutes and repeated every 3 weeks until disease progression or unacceptable toxicity.

SUMMARY:
Patients with metastatic breast cancer with at least 2 brain metastases will receive pembrolizumab every 3 weeks. Patients will undergo stereotactic radiosurgery (SRS) to one of the brain lesions. Pembrolizumab infusion will be given on Day 4 (+/-1) after SRS treatment at the standard dose of 200mg IV over 30 minutes and repeated every 3 weeks until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Patients with metastatic breast cancer with at least 2 brain metastases, eligible to receive SRS. Patients will complete radiation therapy within 1 week and Pembrolizumab may be continued every 3 weeks until evidence of brain progression or serious adverse toxicity. Patients will be followed until death.

Pembrolizumab infusion will be given on Day 4 (+/-1) after SRS treatment at the standard dose of 200mg IV over 30 minutes and repeated every 3 weeks until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Neurological function status 0, 1, 2
* Men and/or pre- or post-menopausal women with metastatic breast cancer with at least 2 intracranial untreated and measurable (≥ 5mm) metastases as visualized on brain MRI
* A diagnostic contrast enhanced MRI demonstrating at least 2 and no more than 10 measurable lesions in the brain, (≥5mm in size), performed within two weeks prior to treatment
* Maximum diameter of treated lesions should be <4cm in size
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document
* Prior SRS is permitted, however the lesions targeted for treatment on trial need to be previously untreated by SRS
* Patients who have undergone prior subtotal resection are eligible providing that residual disease is <4cm in maximum diameter: the cavity will be treated as - - - Continuing a concurrent use of hormonal therapy or anti-Her2 neu therapy is allowed, if the patient exhibits brain metastases progression during these treatments
* Enrolled patients should have a two-week washout period from last systemic treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Contraception duration of 120 days
* Adequate bone marrow reserve and liver function

Exclusion Criteria:

* Active connective tissue disorders, such as lupus or scleroderma requiring flare therapy
* Patients who have undergone complete resection of all known brain metastases
* Inability to obtain histologic proof of breast cancer
* Target lesion metastasis within 5mm of the optic apparatus so that some portion of the optic nerve or chiasm would be included in the SRS field
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy (second primary) that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy..Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with metastatic breast cancer
Enrollment: 41 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response for non-irradiated brain lesions at 8 weeks according to RECIST1.1 | 8 weeks
  detect abscopal responses in non-irradiated brain metastases, followed at routine post SRS brain MRI (evaluated at 8 weeks post-treatment, +/- one week) according to Response Evaluation criteria in Solid Tumors (RECIST1.1)
Correlation of abscopal responses with the radiation dose received | 1 year
  Correlate potential abscopal responses with their radiation dose exposure
Overall survival - assessed from the start of study drug until death in non-irradiation metastases in the rest of the body by routine imaging. | 3 years
  detect systemic objective responses in non-irradiated metastases in the rest of the body, by routine imaging

SECONDARY OUTCOMES:
Number of participants with abscopal response will be assessed. | up to 12 weeks
  Evaluation of an abscopal effect elsewhere in the body. This will be assessed by serial CT based imaging performed every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No